CLINICAL TRIAL: NCT04757480
Title: Ultrasound Guided Thoracolumbar Interfascial Plane Block Versus Bilateral Ultrasound Guided Erector Spinae Plane Block for Post-Operative Pain Management In Lumbar Laminectomy
Brief Title: Thoracolumbar Interfascial Plane Block Versus Bilateral Erector Spinae Plane Block In Lumbar Laminectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aliaa Mohammad Abdel Reeheem Abdel kader, Assistant lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33444/10/19
Record Dates: First submitted 2021-02-14; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain; Lumbar Laminectomy; Thoracolumbar Interfascial Plane Block; Erector Spinae Plane Block; Ultrasound
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracolumbar Interfascial Plane Block (TLIP) (Experimental)
  Interventions: Procedure: Thoracolumbar Interfascial Plane Block (TLIP)
- Bilateral Erector Spinae plane Block (ESB) (Experimental)
  Interventions: Procedure: Bilateral Erector Spinae plane Block (ESB)

INTERVENTIONS:
Procedure: Thoracolumbar Interfascial Plane Block (TLIP) — (20ml) (plain bupivacaine 0.25% on each side toward the LG-MF interface.
  Arms: Thoracolumbar Interfascial Plane Block (TLIP)
Procedure: Bilateral Erector Spinae plane Block (ESB) — Will receive (20ml) (plain bupivacaine 0.25% injected beneath the erector spinae muscle sheath) at the level of the eighth thoracic segment (T8).
  Arms: Bilateral Erector Spinae plane Block (ESB)

SUMMARY:
The aim of this prospective randomized trial is to compare the efficacy ultrasound guided thoracolumbar interfascial plane block versus bilateral ultrasound guided erector spinae plane block for post-operative pain management after lumbar laminectomy

ELIGIBILITY:
Inclusion Criteria:

* Seventy cases with herniated lumbar disc scheduled for lumbar single-level or multiple-level lumbar discectomy with American Society of Anesthesiologists physical status (ASA) I or II aged between 21 and 60 years of both genders.

Exclusion Criteria:

1. Body mass index >32
2. History of relevant allergy to any of the drugs used in the procedure
3. Previous lumbar spine surgery or back surgery with planed spinal fixation

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
Degree of pain by visual Analog Scale (VAS) score at rest | First 24 hours postoperative
  Pain scores will be observed and recorded using the Visual Analog Scale (VAS) both at rest and during movement. The scores will be recorded in the ward at 2, 4, 8, 12, and 24 h.
  VAS score from 0 to 10 (0: No pain, 10: The worst pain)

SECONDARY OUTCOMES:
Degree of pain by visual Analog Scale (VAS) score at movement | First 24 hours postoperative
  Pain scores will be observed and recorded using the Visual Analog Scale (VAS) both at rest and during movement. The scores will be recorded in the ward at 2, 4, 8, 12, and 24 h VAS score from 0 to 10 (0: No pain, 10: The worst pain)
Total rescue analgesics consumption | First 24 hours postoperative
The time to first analgesic | First 24 hours postoperative
24-h morphine consumption | First 24 hours postoperative
Side effects associated with morphine | First 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available with reasonalble consent
Supporting Information: Study Protocol, SAP